CLINICAL TRIAL: NCT00002059
Title: A Double-Blind Placebo Controlled Study To Determine the Optimal Immunopharmacological Dose Level of Isoprinosine in Immunodepressed Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newport Pharmaceuticals International (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 008E; ISO-133-USA
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1989-06

CONDITIONS: HIV Infections
Keywords: T-Lymphocytes, Suppressor-Effector; Neoplasms; Inosine Pranobex; Killer Cells; T-Lymphocytes, Helper-Inducer; Acquired Immunodeficiency Syndrome; AIDS-Related Complex
MeSH Terms: conditions — HIV Infections; Neoplasms; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Inosine Pranobex

INTERVENTIONS:
Drug: Inosine pranobex

SUMMARY:
The objective of this double-blind placebo-controlled study is to evaluate the effect of Isoprinosine in a group of homogenous male volunteers who present with immunologic defects relative to:

* Comparison of total helper and suppressor T-cell number between the groups.
* Comparison of the phytohemagglutinins (PHA) and concanavalin A lymphoproliferative response and natural killer (NK) cell activity between the groups.
* Determination of the clinical course of the volunteers after discontinuance of Isoprinosine.

ELIGIBILITY:
Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Opportunistic infections or Kaposi's sarcoma.
* Critical illness.
* History of gout, urolithiasis, nephrolithiasis, renal dysfunction, and severe gastric ulcer.

Concurrent Medication:

Excluded:

* Steroids.
* Cytotoxic immunosuppressive agents.

Concurrent Treatment:

Excluded:

* Radiotherapy.

The following are excluded:

* Opportunistic infections or Kaposi's sarcoma.
* Critically ill patients.
* Patients receiving steroids, cytotoxic immunosuppressive agents, and/or radiotherapy.
* Patients who have received any other immunotherapy.
* Patients with a history of gout, urolithiasis, nephrolithiasis, renal dysfunction, and severe gastric ulcer.

Prior Medication:

Excluded:

* Any other immunotherapy.

Patients who fall into the group which is at risk of developing cutaneous sarcoma and/or opportunistic diseases but at present have no signs or symptoms of these diseases.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Newport Pharmaceuticals International Inc, Laguna Hills, California, United States